CLINICAL TRIAL: NCT02212470
Title: Randomized Controlled Trial of Paclitaxel Drug-coated Balloons vs. Nitinol Stent for Femoropopliteal Obstructions - The PAVENST Trial
Brief Title: Drug Eluting Balloon Angioplasty Versus Nitinol Stent Implantation in the Superficial Femoral Artery
Acronym: PAVENST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Fabio H Rossi, MD, PHD, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDPC_3 2014
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Peripheral Arterial Disease; Arterial Occlusive Diseases; Atherosclerosis; Arteriosclerosis; Cardiovascular Diseases; Peripheral Vascular Diseases; Paclitaxel; Plaque, Atherosclerotic; Critical Limb Ischemia
Keywords: Artery; Atherosclerosis; Peripheral; Arterial; Plaque; PTA; Angioplasty; Femoropopliteal; Self Expandable Nitinol Stents
MeSH Terms: conditions — Peripheral Arterial Disease; Arterial Occlusive Diseases; Atherosclerosis; Arteriosclerosis; Cardiovascular Diseases; Peripheral Vascular Diseases; Plaque, Atherosclerotic; Chronic Limb-Threatening Ischemia; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-center, single-blind, non-inferiority, clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Eluting Balloon (Active Comparator): Admiral In.Pact Drug Eluting Balloon
  Interventions: Device: Drug Eluting Balloon Angioplasty
- Nitinol Stent (Active Comparator): Complete SE Self-expandible Nitinol stent
  Interventions: Device: Nitinol stenting

INTERVENTIONS:
Device: Drug Eluting Balloon Angioplasty — Angioplasty with Drug eluting balloon after pre dilatation
  Other Names: Medtronic; Admiral In.Pact
  Arms: Drug Eluting Balloon
Device: Nitinol stenting — Nitinol stent deployment
  Other Names: Medtronic; Complete SE
  Arms: Nitinol Stent

SUMMARY:
The purpose of this study is to evaluate whether the results of drug eluting balloon are non-inferior to the Nitinol stent implantation in the femoropopliteal segment.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years with critical lower limb ischemia,
* Ruhtherford 3 or higher,
* with angiographic documentation of greater than 70% or occlusion in the superficial femoral artery,
* with a maximum extension of 10 cm stenosis.
* The popliteal artery and at least one leg artery must be patent.

Exclusion Criteria:

* Pregnancy,
* thrombophilia,
* coagulation disorders,
* presence of active or recent bleeding,
* severe allergy to iodinated contrast,
* renal or hepatic disease,
* acute limb ischemia,
* prior surgical bypass or angioplasty (with or without stent) on the target artery,
* obstructive disease (stenosis> 50%) of the aortoiliac segment ipsilateral to the target (if the aortoiliac is pre-treated, the patient may be included)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Primary patency | 12 months
  Evaluations will be conducted after 3, 6 and 12 months of the procedure. The ultrasonographic evaluation of the degree of stenosis will use the Systolic Velocity Index (division of the velocity of flow at the point of greatest stenosis by the velocity of flow in normal prior segment). Rates higher than 2.4 indicate stenosis greater than 50%

SECONDARY OUTCOMES:
Rutherford classification | 12 months
  Change in classification from Rutherford evaluated in 3, 6 and 12 months.
Ankle braquial Index | 12 months
  Change in the Ankle braquial Index evaluated in 3, 6 and 12 months
Target Lesion Revascularization | 12 months
  Target Lesion Revascularization rate evaluated in 3, 6 and 12 months
Stent fracture | 12 months
  Stent fracture rate evaluated in 3, 6 and 12 months
Amputation | 12 months
  Major amputation defined as amputation that requires prosthesis
Acute myocardial infarct | 12 months
  Acute myocardial infarct rate evaluated in 3, 6 and 12 months
Death | 12 months
  Death rate evaluated in 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: BRUNO L ALMEIDA, MD, Principal Investigator — Instituto Dante Pazzanese de Cardiologia; FABIO H ROSSI, MD, PHD, Study Director — Instituto Dante Pazzanese de Cardiologia
Locations (1):
- Instituto Dante Pazzanese de Cardiologia, São Paulo, Brazil

REFERENCES:
- [Background] Schillinger M, Sabeti S, Dick P, Amighi J, Mlekusch W, Schlager O, Loewe C, Cejna M, Lammer J, Minar E. Sustained benefit at 2 years of primary femoropopliteal stenting compared with balloon angioplasty with optional stenting. Circulation. 2007 May 29;115(21):2745-9. doi: 10.1161/CIRCULATIONAHA.107.688341. Epub 2007 May 14. PMID 17502568
- [Background] Bosiers M, Torsello G, Gissler HM, Ruef J, Muller-Hulsbeck S, Jahnke T, Peeters P, Daenens K, Lammer J, Schroe H, Mathias K, Koppensteiner R, Vermassen F, Scheinert D. Nitinol stent implantation in long superficial femoral artery lesions: 12-month results of the DURABILITY I study. J Endovasc Ther. 2009 Jun;16(3):261-9. doi: 10.1583/08-2676.1. PMID 19642788
- [Background] Dick P, Wallner H, Sabeti S, Loewe C, Mlekusch W, Lammer J, Koppensteiner R, Minar E, Schillinger M. Balloon angioplasty versus stenting with nitinol stents in intermediate length superficial femoral artery lesions. Catheter Cardiovasc Interv. 2009 Dec 1;74(7):1090-5. doi: 10.1002/ccd.22128. PMID 19859954
- [Background] Laird JR, Katzen BT, Scheinert D, Lammer J, Carpenter J, Buchbinder M, Dave R, Ansel G, Lansky A, Cristea E, Collins TJ, Goldstein J, Cao AY, Jaff MR; RESILIENT Investigators. Nitinol stent implantation vs. balloon angioplasty for lesions in the superficial femoral and proximal popliteal arteries of patients with claudication: three-year follow-up from the RESILIENT randomized trial. J Endovasc Ther. 2012 Feb;19(1):1-9. doi: 10.1583/11-3627.1. PMID 22313193
- [Background] Kawamura Y, Ishii H, Aoyama T, Tanaka M, Takahashi H, Kumada Y, Toriyama T, Murohara T. Nitinol stenting improves primary patency of the superficial femoral artery after percutaneous transluminal angioplasty in hemodialysis patients: a propensity-matched analysis. J Vasc Surg. 2009 Nov;50(5):1057-62. doi: 10.1016/j.jvs.2009.07.017. Epub 2009 Sep 26. PMID 19782527
- [Background] Nguyen BN, Conrad MF, Guest JM, Hackney L, Patel VI, Kwolek CJ, Cambria RP. Late outcomes of balloon angioplasty and angioplasty with selective stenting for superficial femoral-popliteal disease are equivalent. J Vasc Surg. 2011 Oct;54(4):1051-1057.e1. doi: 10.1016/j.jvs.2011.03.283. Epub 2011 Jun 2. PMID 21636240
- [Background] Kasapis C, Henke PK, Chetcuti SJ, Koenig GC, Rectenwald JE, Krishnamurthy VN, Grossman PM, Gurm HS. Routine stent implantation vs. percutaneous transluminal angioplasty in femoropopliteal artery disease: a meta-analysis of randomized controlled trials. Eur Heart J. 2009 Jan;30(1):44-55. doi: 10.1093/eurheartj/ehn514. Epub 2008 Nov 21. PMID 19028778
- [Background] Mwipatayi BP, Hockings A, Hofmann M, Garbowski M, Sieunarine K. Balloon angioplasty compared with stenting for treatment of femoropopliteal occlusive disease: a meta-analysis. J Vasc Surg. 2008 Feb;47(2):461-9. doi: 10.1016/j.jvs.2007.07.059. Epub 2007 Oct 22. PMID 17950563
- [Background] Krankenberg H, Schluter M, Steinkamp HJ, Burgelin K, Scheinert D, Schulte KL, Minar E, Peeters P, Bosiers M, Tepe G, Reimers B, Mahler F, Tubler T, Zeller T. Nitinol stent implantation versus percutaneous transluminal angioplasty in superficial femoral artery lesions up to 10 cm in length: the femoral artery stenting trial (FAST). Circulation. 2007 Jul 17;116(3):285-92. doi: 10.1161/CIRCULATIONAHA.107.689141. Epub 2007 Jun 25. PMID 17592075
- [Background] Serruys PW, Kutryk MJ, Ong AT. Coronary-artery stents. N Engl J Med. 2006 Feb 2;354(5):483-95. doi: 10.1056/NEJMra051091. No abstract available. PMID 16452560
- [Background] Lammer J, Bosiers M, Zeller T, Schillinger M, Boone E, Zaugg MJ, Verta P, Peng L, Gao X, Schwartz LB. First clinical trial of nitinol self-expanding everolimus-eluting stent implantation for peripheral arterial occlusive disease. J Vasc Surg. 2011 Aug;54(2):394-401. doi: 10.1016/j.jvs.2011.01.047. Epub 2011 Jun 12. PMID 21658885
- [Background] Dake MD, Scheinert D, Tepe G, Tessarek J, Fanelli F, Bosiers M, Ruhlmann C, Kavteladze Z, Lottes AE, Ragheb AO, Zeller T; Zilver PTX Single-Arm Study Investigators. Nitinol stents with polymer-free paclitaxel coating for lesions in the superficial femoral and popliteal arteries above the knee: twelve-month safety and effectiveness results from the Zilver PTX single-arm clinical study. J Endovasc Ther. 2011 Oct;18(5):613-23. doi: 10.1583/11-3560.1. PMID 21992630
- [Background] Duda SH, Bosiers M, Lammer J, Scheinert D, Zeller T, Tielbeek A, Anderson J, Wiesinger B, Tepe G, Lansky A, Mudde C, Tielemans H, Beregi JP. Sirolimus-eluting versus bare nitinol stent for obstructive superficial femoral artery disease: the SIROCCO II trial. J Vasc Interv Radiol. 2005 Mar;16(3):331-8. doi: 10.1097/01.RVI.0000151260.74519.CA. PMID 15758128
- [Background] Duda SH, Bosiers M, Lammer J, Scheinert D, Zeller T, Oliva V, Tielbeek A, Anderson J, Wiesinger B, Tepe G, Lansky A, Jaff MR, Mudde C, Tielemans H, Beregi JP. Drug-eluting and bare nitinol stents for the treatment of atherosclerotic lesions in the superficial femoral artery: long-term results from the SIROCCO trial. J Endovasc Ther. 2006 Dec;13(6):701-10. doi: 10.1583/05-1704.1. PMID 17154704
- [Background] Werk M, Langner S, Reinkensmeier B, Boettcher HF, Tepe G, Dietz U, Hosten N, Hamm B, Speck U, Ricke J. Inhibition of restenosis in femoropopliteal arteries: paclitaxel-coated versus uncoated balloon: femoral paclitaxel randomized pilot trial. Circulation. 2008 Sep 23;118(13):1358-65. doi: 10.1161/CIRCULATIONAHA.107.735985. Epub 2008 Sep 8. PMID 18779447
- [Background] Micari A, Cioppa A, Vadala G, Castriota F, Liso A, Marchese A, Grattoni C, Pantaleo P, Cremonesi A, Rubino P, Biamino G. Clinical evaluation of a paclitaxel-eluting balloon for treatment of femoropopliteal arterial disease: 12-month results from a multicenter Italian registry. JACC Cardiovasc Interv. 2012 Mar;5(3):331-8. doi: 10.1016/j.jcin.2011.11.010. PMID 22440500
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598
- [Background] Rocha-Singh KJ, Jaff MR, Crabtree TR, Bloch DA, Ansel G; VIVA Physicians, Inc. Performance goals and endpoint assessments for clinical trials of femoropopliteal bare nitinol stents in patients with symptomatic peripheral arterial disease. Catheter Cardiovasc Interv. 2007 May 1;69(6):910-9. doi: 10.1002/ccd.21104. PMID 17377972
- [Background] Leiner T, Kessels AG, Nelemans PJ, Vasbinder GB, de Haan MW, Kitslaar PE, Ho KY, Tordoir JH, van Engelshoven JM. Peripheral arterial disease: comparison of color duplex US and contrast-enhanced MR angiography for diagnosis. Radiology. 2005 May;235(2):699-708. doi: 10.1148/radiol.2352040089. PMID 15858107
- [Background] Freyhardt P, Zeller T, Kroncke TJ, Schwarzwaelder U, Schreiter NF, Stiepani H, Sixt S, Rastan A, Werk M. Plasma levels following application of paclitaxel-coated balloon catheters in patients with stenotic or occluded femoropopliteal arteries. Rofo. 2011 May;183(5):448-55. doi: 10.1055/s-0029-1246028. Epub 2011 Jan 27. PMID 21274828
- [Background] Geiger MA, Guillaumon AT. Primary stenting for femoropopliteal peripheral arterial disease: analysis up to 24 months. J Vasc Bras. 2019 Jan 30;18:e20160104. doi: 10.1590/1677-5449.010416. eCollection 2019. PMID 31191625
- [Background] Krishnan P, Faries P, Niazi K, Jain A, Sachar R, Bachinsky WB, Cardenas J, Werner M, Brodmann M, Mustapha JA, Mena-Hurtado C, Jaff MR, Holden AH, Lyden SP. Stellarex Drug-Coated Balloon for Treatment of Femoropopliteal Disease: Twelve-Month Outcomes From the Randomized ILLUMENATE Pivotal and Pharmacokinetic Studies. Circulation. 2017 Sep 19;136(12):1102-1113. doi: 10.1161/CIRCULATIONAHA.117.028893. Epub 2017 Jul 20. PMID 28729250
- [Background] Schroeder H, Werner M, Meyer DR, Reimer P, Kruger K, Jaff MR, Brodmann M; ILLUMENATE EU RCT Investigators. Low-Dose Paclitaxel-Coated Versus Uncoated Percutaneous Transluminal Balloon Angioplasty for Femoropopliteal Peripheral Artery Disease: One-Year Results of the ILLUMENATE European Randomized Clinical Trial (Randomized Trial of a Novel Paclitaxel-Coated Percutaneous Angioplasty Balloon). Circulation. 2017 Jun 6;135(23):2227-2236. doi: 10.1161/CIRCULATIONAHA.116.026493. Epub 2017 Apr 19. PMID 28424223
- [Background] Schneider PA, Laird JR, Tepe G, Brodmann M, Zeller T, Scheinert D, Metzger C, Micari A, Sachar R, Jaff MR, Wang H, Hasenbank MS, Krishnan P; IN.PACT SFA Trial Investigators. Treatment Effect of Drug-Coated Balloons Is Durable to 3 Years in the Femoropopliteal Arteries: Long-Term Results of the IN.PACT SFA Randomized Trial. Circ Cardiovasc Interv. 2018 Jan;11(1):e005891. doi: 10.1161/CIRCINTERVENTIONS.117.005891. PMID 29326153
- [Result] Iida O, Soga Y, Hirano K, Suzuki K, Yokoi H, Nobuyoshi M, Muramatsu T, Inoue N, Nanto S, Uematsu M. Long-term outcomes and risk stratification of patency following nitinol stenting in the femoropopliteal segment: retrospective multicenter analysis. J Endovasc Ther. 2011 Dec;18(6):753-61. doi: 10.1583/11-3581.1. PMID 22149222
- [Result] Tomoi Y, Soga Y, Takahara M, Fujihara M, Iida O, Kawasaki D, Ando K. Spot stenting versus full coverage stenting after endovascular therapy for femoropopliteal artery lesions. J Vasc Surg. 2019 Oct;70(4):1166-1176. doi: 10.1016/j.jvs.2018.12.044. Epub 2019 Mar 6. PMID 30850285
- [Result] Abdoli S, Mert M, Lee WM, Ochoa CJ, Katz SG. Network meta-analysis of drug-coated balloon angioplasty versus primary nitinol stenting for femoropopliteal atherosclerotic disease. J Vasc Surg. 2021 May;73(5):1802-1810.e4. doi: 10.1016/j.jvs.2020.10.075. Epub 2020 Nov 26. PMID 33249205